CLINICAL TRIAL: NCT03394001
Title: Wound Infiltration With Ketorolac Versus Lidocaine for Postoperative Analgesia After Total Abdominal Hysterectomy: a Prospective, Randomized, Double-blind Study.
Brief Title: Wound Infiltration With Ketorolac Versus Lidocaine for Postoperative Analgesia After Total Abdominal Hysterectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwa Mostafa Mohamed Ali Mowafi, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU R47/2017
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Anesthesia
MeSH Terms: interventions — Lidocaine; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine Hydrochloride (Active Comparator): Wound infiltration with Lidocaine
  Interventions: Procedure: Wound infiltration; Drug: Lidocaine Hydrochloride
- Ketorolac tromethamine (Active Comparator): Wound infiltration with Ketorolac
  Interventions: Procedure: Wound infiltration; Drug: Ketorolac tromethamine

INTERVENTIONS:
Procedure: Wound infiltration — Before skin closure,the subcutaneous tissue and skin all around the wound will be infiltrated by 20 mL of the drug then closure of the skin will be done.
Drug: Lidocaine Hydrochloride — 20 ml of 1% Lidocaine solution
  Other Names: Lidocaine Hydrochloride; Lidocaine HCL 50mg/5 ml
  Arms: Lidocaine Hydrochloride
Drug: Ketorolac tromethamine — 20 mL of saline with 30 mg ketorolac
  Other Names: Adolor; Ketorolac tromethamine 30mg/2ml
  Arms: Ketorolac tromethamine

SUMMARY:
The main goal of this study is to compare wound infiltration with ketorolac versus lidocaine for postoperative analgesia in total abdominal hystrectomy (TAH) operation.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and II
* Planned for elective TAH with a Pfannenstiel incision

Exclusion Criteria:

Patients with the following criteria will be excluded from the study;

* ASA physical status more than II
* Body mass index (BMI)>35 kg/m2
* Previous abdominal surgeries
* Malignancy
* Individuals with chronic pain
* A history of severe systemic disease
* A pre-existing neurological or psychiatric illness
* Known to be addict on alcohol or drugs
* Known allergy to the study drugs

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Rescue analgesia time | First 24 hours postoperatively
  Time for first analgesia requirement

SECONDARY OUTCOMES:
Patient's pain score | First 24 hours postoperatively
  Pain score will be done by visual analog scale (VAS) (minimum 0 = no pain, while maximum 10 cm = worst possible pain). Pain score will be recorded just after extubation (taken as 0 h) and after 1, 2, 4, 6, 12, 18 and 24 h later. Patients will be instructed about the usage of VAS scalebefore the operation.
The total analgesic consumption | First 24 hours postoperatively
  Postoperative analgesia will be provided with intramuscular (IM) meperidine 50 mg to both groups when the VAS score is ≥4. The total meperidine consumption will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided